CLINICAL TRIAL: NCT04433429
Title: Lipid Profile and Vascular Remodelling in Young Dyslipidemic Subjects Treated With Nutraceuticals Derived From Red Yeast Rice.
Brief Title: Nutraceuticals and Vascular Remodelling
Acronym: MALTRO
Status: Completed | Type: Observational
Sponsor: Marcello Rattazzi (Other)
Responsible Party: Sponsor-Investigator, Marcello Rattazzi, Associate Professor, University of Padova
Organization: University of Padova (Other)
Other Study IDs: 3497/AO/15
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hypercholesterolemia
Keywords: Atherosclerosis; Carotid; Lipid profile
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RYR plus CoQ: 333 mg of red yeast rice (RYR, equivalent to 10 mg of Monacolin K) plus 30 mg of Coenzyme Q10 (CoQ10) in a single pill once daily
  Interventions: Dietary Supplement: Liposcudil Plus

INTERVENTIONS:
Dietary Supplement: Liposcudil Plus

SUMMARY:
Aim of the study is to assess the effect of a long-term nutraceutical multitarget approach on lipid profile, inflammatory mediators and vascular remodeling in primary cardiovascular prevention in a setting of controlled dietary habits. The nutraceutical combination used in this study consists of a single pill containing 333 mg of RYR, equivalent to 10 mg of Monacolin K, and 30 mg of Coenzyme Q10 (CoQ10).

ELIGIBILITY:
Inclusion Criteria:

* Total Cholesterol > 150 mg/dl and < 250 mg/dl;
* Triglycerides > 150 mg/dl and < 500 mg/dl;
* Fasting glucose < 126 mg/dl;
* Stable antihypertensive treatment (at least for 6 months) in presence of hypertension.

Exclusion Criteria:

* Total Cholesterol > 250 mg/dl
* Triglycerides > 500 mg/dl
* Previous statin therapy (last 6 months);
* Treatment with hypoglycemic agents and/or fasting glucose > 126 mg/dl;
* Chronic gastrointestinal disorders;
* Chronic kidney disease (eGFR < 60 ml/min/1.73 m2);
* Concomitant treatment with drugs potentially interfering with glucose and lipid metabolism; - History of cardiovascular diseases;
* Proven intolerance to any component of the nutraceutical product;
* Pregnancy or breastfeeding.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with mild hypercholeterolemia and low-to moderate cardiovascular risk profile
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in cholesterol levels at one year | Baseline and one year
  Total Cholesterol will be measured in the blood sample from each patient and expressed as mg/dl
Change from baseline in carotid intima media thickening at one year | Baseline and one year
  Carotid ultrasound examination is performed at baseline and after one year to measure intima-media thickness (IMT). IMT is defined as the distance in mm between the lumen-intima and the media-adventitia interfaces, it is measured at end diastole in the far wall of the right and left sides of the common carotid artery, the bulb and the internal carotid artery. Carotid IMT measurements are expressed as cumulative mean of mean-IMT (m-IMT) recorded in each vascular segment .

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No